CLINICAL TRIAL: NCT01304706
Title: Fluocinolone Acetonide in Diabetic Macular Edema (FAME) Extension Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alimera Sciences (Industry)
Responsible Party: Sponsor
Organization: ANI Pharmaceuticals (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-01-11-008
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Results first posted 2015-05-04 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Fluocinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fluocinolone Acetonide (Experimental)
  Interventions: Drug: Fluocinolone Acetonide

INTERVENTIONS:
Drug: Fluocinolone Acetonide — 0.2 μg/day

SUMMARY:
This study will assess the safety and utility of the new inserter for the administration of ILUVIEN in subjects with diabetic macular edema.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who previously participated in the FAME studies and subjects with chronic DME considered insufficiently responsive to available therapies.
2. In the judgment of the Investigator, the subject will benefit from treatment with ILUVIEN.
3. Ability and willingness to comply with the treatment and follow up procedures.
4. Ability to understand and sign the Informed Consent Form. No expectation that subject will be moving out of the area of the clinical center to an area not covered by another clinical center during the next 12 months.

Exclusion Criteria:

1. Pregnant, lactating females or females of childbearing potential (unless using reliable contraception, i.e. double barrier, surgical sterilization, oral contraceptives, Norplant, intrauterine device (IUD)
2. Glaucoma, defined as glaucomatous anatomical changes of the optic disc and/or visual field changes at screening in the study eye
3. Retinal or choroidal neovascularization due to ocular conditions other than diabetic retinopathy (e.g., presumed ocular histoplasmosis, high myopia (spherical equivalent > 8 diopters), macular degeneration)
4. Any active viral, fungal or bacterial disease of the cornea or conjunctiva or any history of a potentially recurrent infection which could be activated by treatment with a steroid, (e.g., ocular herpes simplex virus)
5. Known or suspected hypersensitivity to any of the ingredients of the investigational product or to other corticosteroids
6. History of uncontrolled IOP elevation with steroid use that did not respond to topical therapy or IOP-lowering procedure
7. History or presence of any disease or condition (malignancy) that in the investigator's opinion would preclude study treatment or follow-up
8. Any lens opacity which significantly impairs vision, in the opinion of the investigator.
9. Peripheral retinal detachment in prospective area of insertion
10. Participation in another clinical trial within 12 weeks before the screening visit or during the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-04; Primary Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Alpharetta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fluocinolone Acetonide
Started | 121
Completed | 104
Not Completed | 17
Not completed — Adverse Event | 2
Not completed — Lack of Efficacy | 1
Not completed — Death | 3
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 7
Not completed — Discontinued due to failed drug admin. | 1

BASELINE CHARACTERISTICS:
Arm/Group | Fluocinolone Acetonide
Number analyzed (Participants) | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (9.29)
Age, Customized [Number; unit: participants]
  <35 | 0
  35-44 | 3
  45-54 | 14
  55-64 | 42
  65-74 | 43
  75-84 | 17
  >=85 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 72
Region of Enrollment [Number; unit: participants]
  United States | 120

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: This is a measurement of the number of subjects who experienced an adverse event and/or a serious adverse event during the trial.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Fluocinolone Acetonide
Number analyzed (Participants) | 120
participants
  Adverse Event | 100
  Serious Adverse Event | 42

ADVERSE EVENTS:
Arm/Group | Fluocinolone Acetonide
Serious Adverse Events (participants affected / at risk) | 42/120
Other Adverse Events (participants affected / at risk) | 100/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluocinolone Acetonide (N=120)
Angina pectoris (Cardiac disorders) | 2 (2)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 4 (4)
Myocardial infarction (Cardiac disorders) | 5 (5)
Ocular hypertension (Eye disorders) | 1 (1) — #Study eye
Retinal detachment (Eye disorders) | 1 (1) — #Fellow eye
Vitreous haemorrhage (Eye disorders) | 1 (1) — #Fellow eye
Oesophagitis (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 2 (2)
Generalised oedema (General disorders) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Intraocular pressure increased (Investigations) | 3 (4) — #Study eye
Gout (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cataract operation (Surgical and medical procedures) | 5 (5) — #Study eye
Cataract operation (Surgical and medical procedures) | 5 (5) — #Fellow eye
Colostomy (Surgical and medical procedures) | 1 (1)
Glaucoma surgery (Surgical and medical procedures) | 2 (2) — #Study eye
Glaucoma surgery (Surgical and medical procedures) | 1 (1) — #Fellow eye
Surgery (Surgical and medical procedures) | 1 (1)
Trabeculectomy (Surgical and medical procedures) | 1 (1) — #Fellow eye
Trabeculoplasty (Surgical and medical procedures) | 1 (1) — #Study eye
Vitrectomy (Surgical and medical procedures) | 5 (5) — #Fellow eye
Hypertension (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluocinolone Acetonide (N=120)
Anaemia (Blood and lymphatic system disorders) | 6 (6)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1)
Aortic valve sclerosis (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Cardiomegaly (Cardiac disorders) | 2 (2)
Coronary artery disease (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Hyperparathyroidism secondary (Endocrine disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 4 (5)
Altered visual depth perception (Eye disorders) | 1 (1) — #Study eye
Blepharitis (Eye disorders) | 3 (3) — #Study eye
Blepharitis (Eye disorders) | 3 (3) — #Fellow eye
Borderline glaucoma (Eye disorders) | 1 (1) — #Study eye
Cataract (Eye disorders) | 12 (15) — #Study eye
Cataract (Eye disorders) | 9 (10) — #Fellow eye
Cataract cortical (Eye disorders) | 1 (1) — #Fellow eye
Cataract nuclear (Eye disorders) | 1 (1) — #Study eye
Cataract nuclear (Eye disorders) | 1 (1) — #Fellow eye
Cataract subcapsular (Eye disorders) | 3 (3) — #Study eye
Cataract subcapsular (Eye disorders) | 2 (2) — #Fellow eye
Conjunctival haemorrhage (Eye disorders) | 28 (28) — #Study eye
Conjunctival haemorrhage (Eye disorders) | 2 (2) — #Fellow eye
Conjunctival hyperaemia (Eye disorders) | 2 (2) — #Study eye
Conjunctivitis (Eye disorders) | 1 (1) — #Study eye
Conjunctivitis (Eye disorders) | 1 (1) — #Fellow eye
Corneal striae (Eye disorders) | 1 (1) — #Study eye
Corneal striae (Eye disorders) | 1 (1) — #Fellow eye
Deposit eye (Eye disorders) | 1 (1) — #Study eye
Diabetic retinal oedema (Eye disorders) | 1 (1) — #Fellow eye
Diabetic retinopathy (Eye disorders) | 1 (1) — #Study eye
Diabetic retinopathy (Eye disorders) | 2 (2) — #Fellow eye
Diplopia (Eye disorders) | 1 (1) — #Study eye
Diplopia (Eye disorders) | 1 (1) — #Fellow eye
Dry eye (Eye disorders) | 5 (5) — #Study eye
Dry eye (Eye disorders) | 3 (3) — #Fellow eye
Erythema of eyelid (Eye disorders) | 1 (1) — #Study eye
Erythema of eyelid (Eye disorders) | 1 (1) — #Fellow eye
Eye discharge (Eye disorders) | 2 (2) — #Study eye
Eye discharge (Eye disorders) | 1 (1) — #Fellow eye
Eye haemorrhage (Eye disorders) | 2 (2) — #Fellow eye
Eye irritation (Eye disorders) | 2 (2) — #Study eye
Eye irritation (Eye disorders) | 1 (1) — #Fellow eye
Eye pain (Eye disorders) | 11 (13) — #Study eye
Eye pruritus (Eye disorders) | 2 (2) — #Study eye
Eye pruritus (Eye disorders) | 2 (2) — #Fellow eye
Eyelid cyst (Eye disorders) | 1 (1) — #Fellow eye
Eyelid oedema (Eye disorders) | 2 (2) — #Study eye
Eyelid ptosis (Eye disorders) | 1 (1) — #Study eye
Eyelid ptosis (Eye disorders) | 1 (1) — #Fellow eye
Eyelids pruritus (Eye disorders) | 1 (1) — #Study eye
Foreign body sensation in eyes (Eye disorders) | 1 (2) — #Study eye
Glaucoma (Eye disorders) | 3 (3) — #Study eye
Glaucoma (Eye disorders) | 1 (1) — #Fellow eye
Halo vision (Eye disorders) | 1 (1) — #Study eye
Iris neovascularisation (Eye disorders) | 1 (1) — #Study eye
Keratitis (Eye disorders) | 1 (1) — #Study eye
Keratitis (Eye disorders) | 1 (1) — #Fellow eye
Lacrimation increased (Eye disorders) | 1 (1) — #Study eye
Macular degeneration (Eye disorders) | 1 (1) — #Fellow eye
Macular hole (Eye disorders) | 1 (1) — #Study eye
Macular oedema (Eye disorders) | 1 (1) — #Fellow eye
Maculopathy (Eye disorders) | 5 (5) — #Study eye
Maculopathy (Eye disorders) | 2 (2) — #Fellow eye
Metamorphopsia (Eye disorders) | 1 (1) — #Study eye
Myodesopsia (Eye disorders) | 6 (7) — #Study eye
Myodesopsia (Eye disorders) | 2 (2) — #Fellow eye
Ocular discomfort (Eye disorders) | 1 (1) — #Study eye
Ocular hyperaemia (Eye disorders) | 5 (5) — #Study eye
Ocular hypertension (Eye disorders) | 7 (9) — #Study eye
Ocular hypertension (Eye disorders) | 1 (1) — #Fellow eye
Open angle glaucoma (Eye disorders) | 1 (1) — #Study eye
Papilloedema (Eye disorders) | 1 (1) — #Fellow eye
Photophobia (Eye disorders) | 4 (4) — #Study eye
Photophobia (Eye disorders) | 1 (1) — #Fellow eye
Photopsia (Eye disorders) | 2 (2) — #Study eye
Posterior capsule opacification (Eye disorders) | 1 (1) — #Study eye
Retinal depigmentation (Eye disorders) | 1 (1) — #Fellow eye
Retinal detachment (Eye disorders) | 1 (1) — #Fellow eye
Retinal exudates (Eye disorders) | 2 (2) — #Study eye
Retinal exudates (Eye disorders) | 3 (3) — #Fellow eye
Retinal haemorrhage (Eye disorders) | 1 (1) — #Study eye
Retinal haemorrhage (Eye disorders) | 3 (3) — #Fellow eye
Retinal pigment epitheliopathy (Eye disorders) | 1 (1) — #Fellow eye
Vision blurred (Eye disorders) | 3 (4) — #Study eye
Visual acuity reduced (Eye disorders) | 6 (6) — #Study eye
Visual acuity reduced (Eye disorders) | 2 (2) — #Fellow eye
Visual impairment (Eye disorders) | 2 (2) — #Study eye
Visual impairment (Eye disorders) | 2 (2) — #Fellow eye
Vitreous detachment (Eye disorders) | 3 (3) — #Study eye
Vitreous detachment (Eye disorders) | 1 (1) — #Fellow eye
Vitreous haemorrhage (Eye disorders) | 8 (8) — #Study eye
Vitreous haemorrhage (Eye disorders) | 5 (7) — #Fellow eye
Vitritis (Eye disorders) | 1 (1) — #Study eye
Abdominal discomfort (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
Gingival disorder (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1) — #Fellow eye
Proctalgia (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Generalised oedema (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 2 (2)
Seasonal allergy (Immune system disorders) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Gastritis viral (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 3 (3)
Genital infection fungal (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Histoplasmosis (Infections and infestations) | 1 (1)
Infected cyst (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 2 (2)
Localised infection (Infections and infestations) | 2 (2)
Osteomyelitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 4 (5)
Tooth abscess (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 6 (6)
Urinary tract infection (Infections and infestations) | 7 (8)
Vaginal infection (Infections and infestations) | 1 (1)
Avulsion fracture (Injury, poisoning and procedural complications) | 1 (1)
Corneal abrasion (Injury, poisoning and procedural complications) | 1 (1) — #Study eye
Excoriation (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 5 (5)
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1)
Blood cholesterol increased (Investigations) | 1 (1)
Blood magnesium decreased (Investigations) | 1 (1)
Blood pressure increased (Investigations) | 1 (1)
Blood triglycerides increased (Investigations) | 1 (1)
Intraocular pressure increased (Investigations) | 13 (15) — #Study eye
Intraocular pressure increased (Investigations) | 3 (3) — #Fellow eye
Intraocular pressure test abnormal (Investigations) | 1 (1) — #Study eye
Platelet count increased (Investigations) | 1 (1)
Red blood cell count decreased (Investigations) | 1 (1)
Very low density lipoprotein increased (Investigations) | 1 (1)
White blood cell count increased (Investigations) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1)
Gout (Metabolism and nutrition disorders) | 2 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Head deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3)
Carpal tunnel syndrome (Nervous system disorders) | 1 (2)
Complex regional pain syndrome (Nervous system disorders) | 1 (1)
Demyelination (Nervous system disorders) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Encephalopathy (Nervous system disorders) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 4 (4)
Hypoaesthesia (Nervous system disorders) | 2 (2)
Neuritis (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 3 (3)
Presyncope (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (2)
Syncope (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 2 (2)
VIth nerve paralysis (Nervous system disorders) | 1 (1)
Visual field defect (Nervous system disorders) | 1 (1) — #Study eye
Visual field defect (Nervous system disorders) | 1 (1) — #Fellow eye
Depression (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 3 (3)
Renal failure chronic (Renal and urinary disorders) | 4 (4)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cutis laxa (Skin and subcutaneous tissue disorders) | 1 (1) — #Study eye
Cutis laxa (Skin and subcutaneous tissue disorders) | 1 (1) — #Fellow eye
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1)
Arterial stenosis limb (Vascular disorders) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 4 (5)
Hypotension (Vascular disorders) | 1 (1)
Leriche syndrome (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days